CLINICAL TRIAL: NCT04068389
Title: Study of the Permeability of Atmospheric Particles Placenta (Fine and Ultrafine Particles): Analysis of Fetal Retention
Brief Title: Ultrafine Particles and Fetal Contamination
Acronym: FOETOPUF
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2008/04
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lung; Premature; Pollution; Exposure
Keywords: Atmospheric particles
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fetal lung samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pulmonary Tissue Collection — Pulmonary Tissue Collection

SUMMARY:
The objective of this study is to evaluate the transplacental passage of fine and ultrafine particles (nanoparticles) inhaled by the mother.

DETAILED DESCRIPTION:
Epidemiological studies have demonstrated the harmful effects of particulate air pollution on the progress of pregnancy and postnatal health.

Experimental studies have suggested the transplacental passage of asbestos fibers, but despite the strong growth in the use and production of fine and ultrafine particles, no study has examined the permeability of the placenta to these compounds or the exposures fetuses that may result.

The objective of this study is to evaluate the transplacental passage of fine and ultrafine particles (nanoparticles) inhaled by the mother.

ELIGIBILITY:
Inclusion Criteria:

- All women volunteers for whom a medical termination of pregnancy is proposed for a fetus older than 22 weeks (weight over 500g).

Exclusion Criteria:

* Refusal of participation of the patient.
* Fetus with malformation syndrome affecting pulmonary perfusion.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnacy women
Study Population: Women with a medical termination of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2009-12-22 (Actual); Primary Completion 2012-11-09 (Actual); Study Completion 2012-11-09 (Actual)

PRIMARY OUTCOMES:
Presence of fine particles in fetal lung samples yes/no | At the screening
  Analysis in electron microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Olivia OCHRYMCZUK, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No